CLINICAL TRIAL: NCT04584268
Title: A Randomized Controlled Trial of a Longitudinal Mindfulness Intervention to Decrease Burnout in Medical Residents
Brief Title: Longitudinal Mindfulness Intervention to Decrease Burnout in Medical Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Prater, Assistant Professor in Medicine and Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201904014
Record Dates: First submitted 2020-07-23; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Burnout
Keywords: burnout; medical residents
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness (Experimental): 3 30 minute in person interventions as well as promotion and involvement of self-guided meditations on the Insight Timer smart phone application
  Interventions: Behavioral: mindfulness
- control (Active Comparator): standard medical resident education
  Interventions: Other: standard medical education

INTERVENTIONS:
Behavioral: mindfulness — in person and smart phone application mindfulness practice
  Arms: mindfulness
Other: standard medical education — standard medical education / control
  Arms: control

SUMMARY:
This was a single-site RCT to assess the effect of a longitudinal mindfulness intervention on burnout for first-year (PGY-1) internal medicine (IM) and pediatrics residents. The primary outcome was Maslach Burnout Inventory MBI) scores at baseline and 12 month follow-up. Secondary outcomes were feasibility and perceived benefit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Washington University (WUSM) first year residents in internal medicine and pediatrics

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory (MBI) | 1 year
  burnout score on MBI (score range 0-132); based on three components: emotional exhaustion, depersonalization, and personal accomplishment)
feasibility of intervention in graduate medical education | 1 year
  ability to insert into the curriculum without barriers or disruption of other education activities, assessed by interviews from residency leadership

SECONDARY OUTCOMES:
evaluation of intervention | 1 year
  survey to assess opinion of intervention (Likert scale)
effect on mindfulness practice | 1 year
  survey question to assess pre and post-intervention frequency of practicing mindfulness

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: protocol and SAP now. CSR upon publication